CLINICAL TRIAL: NCT05835726
Title: Daratumumab-containing Induction Effects on Stem Cells Mobilization, colLection and Engraftment in Newly Diagnosed Multiple MyelomA Patients (DILEMMA).
Brief Title: Daratumumab-containing Induction Effects on Stem Cells Mobilization, colLection and Engraftment in Newly Diagnosed Multiple MyelomA Patients.
Acronym: DILEMMA
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5446
Record Dates: First submitted 2023-04-19; First posted 2023-04-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma; Daratumumab; Autologous Stem Cell Transplantation; Leukapheresis
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases (prospective cohort): Patients who fulfill the inclusion criteria (newly diagnosed multiple myeloma patients undergoing daratumumab-containing induction regimens).
  Interventions: Drug: Daratumumab
- Controls: Patients with newly diagnosed multiple myeloma who received standard VTD (VTD:bortezomib-thalidomide and dexamethasone) induction, subsequent stem cell mobilization, and tandem autologous stem cell transplant before the introduction of daratumumab in our local practice from January 2020 to December 2021.

INTERVENTIONS:
Drug: Daratumumab — NDMM (newly diagnosed multiple myeloma) who fulfill the inclusion criteria, candidate to stem cell mobilization, collection, and autologous stem cell transplant who receive a Daratumumab-containing induction regimen.
  Other Names: Darzalex
  Groups: Cases (prospective cohort)

SUMMARY:
Daratumumab is a human first-in-class monoclonal antibody that targets a cluster of differentiation (CD) 38, a cell surface protein that is overexpressed on multiple myeloma (MM) cells, showing significant activity in relapsed/refractory disease. More recently, it was demonstrated that the addition of daratumumab to pre-autologous hematopoietic stem cell transplant (ASCT) induction regimens in newly diagnosed multiple myeloma increased the rate of complete responses and disease-free survival. However, in consideration of the expression of CD38 antigen also by stem cells, daratumumab could exert effects on their mobilization, collection, and engraftment. The primary objective of this retrospective/prospective observational study is to investigate the impact of adding daratumumab to standard induction regimens (VTD:bortezomib-thalidomide and dexamethasone, VD: bortezomib and dexamethasone) on stem cell mobilization in patients with newly diagnosed multiple myeloma (NDMM) who are candidates for ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* NDMM candidate to stem cell mobilization, collection, and ASCT who received a Daratumumab-containing induction regimen.
* Signed written informed consent to study participation.

Exclusion Criteria:

* Age <18 y.o.
* Inability to obtain written informed consent.
* Patients not proceeding to stem cell mobilization because of disease progression.
* Patients not eligible for high-dose cyclophosphamide according to baseline cardiologic evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases (prospective cohort): Patients with newly diagnosed multiple myeloma candidate to stem cell mobilization, collection, and autologous stem cell transplant who receive a Daratumumab-containing induction regimen.
  Controls: Patients with newly diagnosed multiple myeloma who received standard VTD induction, subsequent stem cell mobilization, and tandem autologous stem cell transplant before the introduction of daratumumab in our local practice from January 2020 to December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
To assess the difference in the mean number of collected CD34+ cells/kg during total harvest between Daratumumab and control group. | 12 months
  To assess the difference in the mean number of collected CD34+ cells/kg during total harvest between Daratumumab and control group.

SECONDARY OUTCOMES:
Proportion (%) of patients achieving at least two minimum transplant doses (4x10^6 CD34+ cells/kg) at first day of apheresis in Daratumumab versus control group. | 12 months
  Proportion (%) of patients achieving at least two minimum transplant doses (4x10^6 CD34+ cells/kg) at first day of apheresis in Daratumumab versus control group.
Proportion (%) of patients who received plerixafor rescue for poor mobilization in Daratumumab versus control group. | 12 months
  Proportion (%) of patients who received plerixafor rescue for poor mobilization in Daratumumab versus control group.
Graft composition in Daratumumab group in term of concentration of CD34+ cells x10^6/kg, TNC (total nucleated cells) x 10^8/kg, and MNC (mononuclear cells) x 10^8/kg. | 12 months
  Graft composition in Daratumumab group in term of concentration of CD34+ cells x10^6/kg, TNC (total nucleated cells) x 10^8/kg, and MNC (mononuclear cells) x 10^8/kg.
Rate (%) of CD38 expression and clonogenic potential of collected CD34+ cells in both groups. | 12 months
  Rate (%) of CD38 expression and clonogenic potential of collected CD34+ cells in both groups.
To compare transplant outcome in term of time (days) to platelets and neutrophils engraftment in Daratumumab versus control group. | 12 months
  To compare transplant outcome in term of time (days) to platelets and neutrophils engraftment in Daratumumab versus control group.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Teofili, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A.Gemelli IRCCS, Rome, Italy